CLINICAL TRIAL: NCT06809049
Title: Music Intervention for Brain-Heart Disease in Myotonic Dystrophy Type 1 (DM1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanns Lochmuller (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor-Investigator, Hanns Lochmuller, Senior Scientist, Children's Hospital of Eastern Ontario
Organization: Children's Hospital of Eastern Ontario (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24/143X; CFREF-2022-00007 (Other Grant/Funding Number: Canada First Research Excellence Fund); BHI 23-118 (Other Grant/Funding Number: uOttawa Brain-Heart Interconnectome)
Record Dates: First submitted 2025-01-27; First posted 2025-02-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Myotonic Dystrophy, Congenital; Myotonic Dystrophy, Type 1 (DM1); Myotonic Dystrophy Type 1; Myotonic Dystrophy Type 1 (DM1)
Keywords: Music intervention; Myotonic dystrophy; DM1; Rare disease; Dalcroze music education
MeSH Terms: conditions — Myotonic Dystrophy; Rare Diseases

STUDY DESIGN:
Intervention Model Description: Participants will be grouped with 5-7 other participants of similar age and ability for the music education sessions. All participants will receive the music intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Music Intervention (Experimental): All participants will receive weekly Dalcroze music education sessions.
  Interventions: Behavioral: Dalcroze music education

INTERVENTIONS:
Behavioral: Dalcroze music education — Dalcroze is a type of music education which focuses on free and improvised movement, as well as structure and choreographed sequences. It has been successfully applied to similar populations as an effective, accessible, and sustainable intervention. We hope to use Dalcroze music education to employ a holistic approach to improve the brain-heart symptoms of children with congenital DM1.

SUMMARY:
The goal of this interventional study is to demonstrate the feasibility and tolerability of Dalcroze music intervention for children with congenital DM1, while providing indications of its effectiveness in improving brain and heart symptoms of DM1. Additionally, information from the collection of biological samples and wearable devices (accelerometer, EEG headband and ECG chest strap) will be used to identify brain-heart biomarkers and outcome measures for use in future research and trials.

Researchers will compare the results of physical and cognitive assessments for each participant to assessments from baseline after 10 weeks of weekly music sessions. Qualitative measures (questionnaires and focus groups) will inform the feasibility of this intervention for this population. The main questions this study aims to answer are:

* Are weekly music education sessions feasible for children with DM1?
* Are weekly music education sessions tolerable for children with DM1?

Participants will:

* Attend 45-minute-long music sessions once weekly for 10 weeks.
* Attend two clinic visits for cognitive and physical assessments.
* Provide blood, saliva, stool and urine samples.
* Use wearable devices both at-home and during music sessions.
* Parents/caregivers of participants will complete questionnaires and participate in three focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 6 to 18 with genetically confirmed congenital or infantile-onset myotonic dystrophy type 1 (DM1).
* Participants willing to stay on stable medication from the day of screening to end of study.

Exclusion Criteria:

* Insufficient English language skills to complete required assessments and questionnaires.
* Participant is non-verbal.
* Failure to provide signed informed consent by participant or designated decision maker (i.e. parent, legal guardian or power of attorney).
* Failure to provide signed informed consent by parents/caregivers for dyad participation.
* Participant is not a resident of Canada, due to risk of attrition.
* Patients for whom - in the opinion of the investigator - it would not be safe to participate in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Attendance to Each Music Session | Over 10-week block of music sessions
  Participant attendance rate to 10 music sessions.
Attendance to Block of Music Sessions | Over 10-week block of music sessions
  The proportion of participants who attend all 10 music sessions.
Qualitative Feedback from Parents/Caregivers Following Each Music Session | Following each music session through to the final music session.
  Parents/Caregivers will complete short questionnaires following each of the 10 music sessions. Questions will focus on recall of participant mood, tiredness and engagement in the 24 hours immediately following each music session.

SECONDARY OUTCOMES:
Change in Physical Performance Assessed by the 6-Minute Walk Test (6MWT) | Baseline and 1 week following the final music session.
  The 6-minute walk test involves the participant walking unaccompanied along a 30m hallway as far as possible within a 6-minute period.
Change from Baseline in Clinical Phenotype Assessed by the Clinician-Completed Congenital DM1 Rating Scale (CDM1-RS) | Baseline and 1 week following the final music session.
  The clinician rates the severity of 11 key symptoms over the past week on a 5-point Likert scale from 0 (least severe) to 4 (most severe).
Change in Global IQ Assessed by Wechsler Abbreviated Scale of Intelligence Second Edition (WASI-II) | Baseline and 1 week following the final music session.
  The WASI-II is a standardized measure of overall intelligence, with a higher score corresponding to higher intellectual ability.
Change in Attention Assessed by Bells Assessment | Baseline and 1 week following the final music session.
  In the Bells assessment, the participant is asked to circle all the bells on a page with other images as distractors. The maximum score is 35/35 bells.
Change in Working Memory Assessed by NIH List Sorting Working Memory Test | Baseline and 1 week following the final music session.
Change in Executive Functioning Assessed by Dimensional Change Card Sort | Baseline and 1 week following the final music session.
  The participant is asked to match a series of picture pairs to a target picture.
Change in Visuospatial Skills Assessed by Rex Complex Figure - Copy | Baseline and 1 week following the final music session.
Change in Episodic Memory Assessed by NIH Picture Sequence Memory Test | Baseline and 1 week following the final music session.
Change in Receptive Vocabulary Assessed by Peabody Picture Vocabulary Test (PPVT-5) | Baseline and 1 week following the final music session.
  A measure of receptive vocabulary with scores ranging from 0 (lower receptive vocabulary skills) to 175 (higher receptive vocabulary skills).
Change in Mood and Anxiety Assessed by Mood and Feelings Questionnaire (MFQ) | Baseline and 1 week following the final music session.
  Participants self-report the applicability of phrases as true, sometimes true, or not true.
Change in Adaptive Functioning Assessed by Vineland Adaptive Behaviour Scale | Baseline and 1 week following the final music session.
Change in Quality of Life Assessed by Pediatric Quality of Life Inventory (PedsQL) | Baseline and 1 week following the final music session.
  Participant and their parents report on the frequency (never to almost always) of specific health-related quality of life problems. A higher score indicates poorer quality of life.
Change in Sleep Quality Assessed by Children's Sleep Habits Questionnaire | Baseline and 1 week following the final music session.
  Parent completed questionnaire to assess participant sleep behaviours. Each question is rate on a 3-point scale. Total scores can range from 33-99, with a score higher than 41 suggesting the presence of a childhood sleep disorder.
Assessment of Cardiac Conduction Defects by Electrocardiogram (ECG) | Baseline and 1 week following the final music session.
  Participants will receive clinical ECG testing to assess for the presence of cardiac conduction defects.
Changes in Attention Assessed by Conners Continuous Performance Test Third Edition (CPT3) | Baseline and 1 week following the final music session.
  Participants are instructed to press the spacebar of a computer each time the letter X appears. A higher score indicates worse performance.
Change in Executive Functioning Assessed by Behaviour Rating Inventory of Executive Functioning (BRIEF2) | Baseline and 1 week following the final music session.
  The score ranges from 80-240, with a higher score indicating greater executive dysfunction.
Change in Physical Performance Assessed by the 10-meter walk/run test (10-mW/RT) | Baseline and 1 week following the final music session.
  For the 10-meter walk/run test, the participant walks/runs without assistance for 12 meters while the time taken to walk from meter 1 to meter 11 is recorded with a stopwatch. The test will be repeated 2-3 times, with a minimum of 10-15 seconds of rest between trials to avoid fatigue.
Change in Physical Activity Assessed by Accelerometer | Baseline and 1 week following the final music session.
  Actigraph wGT3X-BT accelerometer will be worn for continuous tracking of activity for two 7-day periods.
Change in Affect Assessed by Positive and Negative Affect Scale - Child (PANAS-C) | Baseline and 1 week following the final music session.
  Participants self-report the frequency each feeling or emotion was experienced on a 5-point Likert scale.
Change in Anxiety Assessed by State-Trait Anxiety Inventory Scale-5 (STAIS-5) | Baseline and 1 week following the final music session
Change in Sleep Quality Assessed by Electroencephalogram (EEG) Headband | Nightly for 7 days at baseline and 1 week following the final music session.
  Participants will wear a Muse-EEG headband overnight. Measures of sleep architecture will inform overall sleep quality.
Assessment of Heart Rate Variability by Wearable Electrocardiogram (ECG) Chest Strap | Over 7-day period at baseline and following final music intervention.
  Participants will wear a Polar H10 ECG chest strap for at-home monitoring of heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified quantitative data including, results of cognitive and physical assessments and wearable device measurements.
Supporting Information: Study Protocol, ICF
Access Criteria: IPD will be stored within the Brain-Heart Collaborative Portal and accessible to qualified researchers with a research plan approved by a data access committee. Supporting information (protocol and informed consent forms) will be available as a publication.